CLINICAL TRIAL: NCT03952975
Title: Optimal Timing for Performing Loop Electrosurgical Excision Procedure According to Different Menstrual Phase: Which is Best?
Brief Title: Optimal Timing for Performing Loop Electrosurgical Excision Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Principal Investigator, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUGLA SKU
Record Dates: First submitted 2019-05-12; First posted 2019-05-16 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Cervical Precancerous Lesions
Keywords: Loop electrosurgical excision procedure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- follicular phase group (Other): The menstrual dates of patients were normalized to a 28-day cycle with the following formula: adjusted day of the menstrual cycle = (14 X day of the cycle at the time of surgery) / (cycle length of the patient - 14). In light of this formula patients were classified into the follicular phase group (defined as <15 adjusted days, group A).
  Interventions: Other: Vaginal bleeding
- luteal phase group (Other): The menstrual dates of patients were normalized to a 28-day cycle with the following formula: adjusted day of the menstrual cycle = (14 X day of the cycle at the time of surgery) / (cycle length of the patient - 14) [14]. In light of this formula, patients were classified into the luteal phase group (defined as ≥15 adjusted days, group B).
  Interventions: Other: Vaginal bleeding

INTERVENTIONS:
Other: Vaginal bleeding — Vaginal bleeding was classified into four categories according to the timing. Intraoperative bleeding (defined as bleeding that occur during the LEEP procedure), early postoperative bleeding (defined as bleeding that occur between end of the LEEP procedure and home discard), late postoperative bleeding (defined as bleeding that occur within two weeks after the home discard, and required hemostatic interventions such as electrocauterization, gauze packing, or cervical suturing, excluding menstrual bleeding), and persistent postoperative bleeding (defined as vaginal bleeding that occurs more than 2 weeks after the procedure with or without required hemostatic interventions, excluding menstrual bleeding).

SUMMARY:
Cervical precancerous lesions (cervical intraepithelial neoplasia) are frequently diagnosed and treated in women of reproductive-aged [1]. Loop electrosurgical excision procedure (LEEP) is the standard surgical treatment in CIN 2 or 3 [1]. This procedure is an inexpensive, easy to learn and provide specimens for pathological examination with the least major surgical morbidity [2].

Although LEEP is a safe procedure, complications such as postoperative bleeding have been reported. These haemorrhages make patients anxious, undergo unnecessary follow-ups, additional procedures to stop bleeding and interfere in patients daily activities. Various interventions have been attempted to prevent and/or reduce perioperative and/or postoperative haemorrhage after LEEP including vasopressiın, tranexamic acid, Monsel's solution, or local hemostats (TochoSil or Tisseel), but have failed to show a definite advantage over routine practice [2-4].

A hormonal variation during the menstrual cycle is known to affect hemostasis [5] and the blood flow of the genital organ [6,7]. A systematic review of the literature through PubMed, OvidSP, Google Scholar, and Scopus identified only one previous investigation of menstrual cycle period affect blood loss during the LEEP procedure. The authors showed that women had less perioperative bleeding during the follicular phase than during the luteal phase [8]. Two retrospective studies have also demonstrated rhinoplasty and mammoplasty caused more bleeding during the luteal phase and menstruation than during the follicular phase [9,10]. In contrast, other retrospective studies have shown no relation between operative blood loss and the menstrual cycle for hysterectomy, myomectomy, and ovarian cystectomy [11-13] To answer this clinically relevant question, the investigators performed a randomized study comparing perioperative and postoperative bleeding between patients underwent LEEP procedure during the follicular or luteal phase of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Women was ≥ 21 years old
2. Women was not pregnant
3. Women were not menstruating or menopausal status
4. Women with the normal regular menstrual cycle (defined as an interval between 21 and 35 days and duration between 3 and 10 days)
5. Women had one of the following indications for LEEP procedure

   1. a histology-proven, persistent, low grade squamous intraepithelial lesions (LGSIL),
   2. a histology-proven high-grade squamous intraepithelial lesions (HGSIL),
   3. discrepancies between cytological reports and colposcopic impressions,
   4. investigation for unsatisfactory colposcopy,
   5. micro invasion or adenocarcinoma in situ on cervical punch biopsy

Exclusion Criteria:

* Women with cervical or vaginal infection,
* Women with the abnormal menstrual cycle,
* Women taking any medication (or injection) such as oral contraceptives, GnRH agonist, medroxyprogesterone acetate, or anticoagulants
* Women with coagulation defect,
* Women with mental incapacity,
* Women with a history of neurologic deficit,
* Women with previous hysterectomy with removal of the cervix,
* Women with a history of cervical cancer

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
mean early postoperative blood loss | 6 hours
  Estimated early postoperative blood loss was calculated using the difference in hematocrit values taken after LEEP procedure and 6 hours after procedure, according to the following formula: Estimated Blood Loss = estimated blood volume X (hematocrit 1 - hematocrit 2)/hematocrit 1, where the estimated blood volume in milliliters = woman's weight in kilograms X 85

SECONDARY OUTCOMES:
mean intraoperative bleeding | During the LEEP procedure
  The volume of intraoperative blood loss was measured by weighing a gauze sponge during the procedure. Because it is important to collect the blood accurately, we used a specially designed operating gauze sponge and an electronic scale to weigh all the material (with a 1-g deviation range). The LEEP procedure was performed ensuring that all blood lost during the procedure was absorbed with gauzes. We took care to clean all the bleeding with gauze obtained during the procedure.
the rate of late postoperative bleeding | bleeding that occur within four weeks after the home dischard
  late postoperative bleeding (defined as bleeding that occur within four weeks after the home dischard, and required hemostatic interventions such as electrocauterization, gause packing, or cervical suturing, excluding menstrual bleeding).

CONTACTS AND LOCATIONS:
Locations (1):
- Kemal Gungorduk, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paraskevaidis E, Davidson EJ, Koliopoulos G, Alamanos Y, Lolis E, Martin-Hirsch P. Bleeding after loop electrosurgical excision procedure performed in either the follicular or luteal phase of the menstrual cycle: a randomized trial. Obstet Gynecol. 2002 Jun;99(6):997-1000. doi: 10.1016/s0029-7844(02)02003-3. PMID 12052589